CLINICAL TRIAL: NCT03390166
Title: A Phase II/III Double Blinded, Randomized, Controlled, Non-inferiority Trial to Evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine, in Healthy Thai Subjects Aged 18-49 Years
Brief Title: Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Influenza Vaccine in Healthy Thai Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Prof., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Tri Fluvac Vaccine phase 2/3
Record Dates: First submitted 2017-07-06; First posted 2018-01-04 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Influenza
Keywords: GPO Tri Fluvac Vaccine; Tri Fluvac vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: non-inferiority double-blinded, randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPO Tri Fluvac vaccine (Active Comparator): 630 volunteers will receive a single dose of the seasonal trivalent inactivated influenza vaccine (consisting of A/Michigan/45/2015 (H1N1)pdm-09-like virus, A/Hong Kong/4801/2014 (H3N2)-like virus, and B/Brisbane/60/2008-like virus) produced by GPO Thailand. To be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Interventions: Biological: GPO Tri Fluvac vaccine
- Licensed Influenza vaccine (Active Comparator): 315 volunteers will receive acLicensed Influenza vaccine (seasonal trivalent inactivated split virion influenza vaccine recommended for Southern Hemisphere in 2017 (consisting of A/Michigan/45/2015 (H1N1)pdm-09-like virus, A/Hong Kong/4801/2014 (H3N2)-like virus, and B/Brisbane/60/2008-like virus) 0.5 mL administered intramuscularly (IM) in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Licensed influenza vaccine

INTERVENTIONS:
Biological: GPO Tri Fluvac vaccine — The vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Arms: GPO Tri Fluvac vaccine
Biological: Licensed influenza vaccine — The comparator licensed influenza vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Arms: Licensed Influenza vaccine

SUMMARY:
The study is aim to evaluate the immunogenicity and safety with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza vaccine

DETAILED DESCRIPTION:
This is a phase II/III, non-inferiority double-blinded, randomized, controlled trial of immunogenicity and safety with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza vaccine).

A total of about 945 healthy Thai male and female adult volunteers 18 through 49 years of age; 630 participants will be randomized to receive the GPO Tri Fluvac and 315 will receive an active comparator (a 2:1 ratio) (inclusion of ~7% lost to follow-up).

Safety will be assessed for all participants through Day 90 after vaccination. Immunogenicity will be assessed in serum samples obtained at baseline and 21 days after vaccination in a subset of at least 586 individuals randomized to study vaccine and 293 active comparator vaccine recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years old on the day of screening, having Thai ID card or equivalent
* Able to read and write in Thai and sign written informed consent form
* Able to attend all scheduled visits and to comply with all trial procedures.
* Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable, under control or unchanged for the past three months. If medication is used to treat the condition, the medication dose must have been stable for at least one month preceding vaccination.
* For female participants:

  * Not breast feeding, non-pregnant (based on negative urine pregnancy test) and no plan to become pregnant up to Day 60.
  * Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than one year must be willing to use effective contraceptive method to prevent pregnancy until Day 60 after vaccination. Effective methods include intrauterine device, hormonal contraceptives (oral, injectable, patch, implant, ring) or double barrier contraceptives (condom or diaphragm with spermicide). Women with credible history of abstinence may be enrolled at the discretion of the investigator

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Hypersensitivity after previous administration of any vaccine.
* Having a history of H1N1, H3N2 or Flu B infection within 3 months preceding enrollment to the trial
* Vaccination against influenza in the past 6 months preceding enrollment to the trial
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 21 visit.
* History of bronchial asthma, chronic lung diseases, chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression < 6 months prior to immunization
* History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. gentamicin or thimerosal)
* History of Guillain-Barré Syndrome.
* Having acute infection with fever > 38 degree Celsius or noninfectious diseases (within 72 hours) preceding enrollment in the trial
* Volunteers who have been taking immunoglobulin products or have had a blood transfusion during past 3 months before the beginning of the trial or planned receipt of such products prior to the Day 21 visit.
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 945 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Prof., Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University,, Bangkok
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An advertising brochure on this study which was approved by the Institutional Review Board (IRB) was distributed to potential participants. Participants who were interested in participating in this study contacted the investigator. An appointment was made to explain the details of the study individually.
Pre-assignment Details: Pre-assignment Details
  A total of 945 participants who met all inclusion criteria and not of the exclusion criteria were enrolled in the study.
Period: Overall Study
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
Started | 630 | 315
Completed | 618 | 305
Not Completed | 12 | 10
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 6 | 4
Not completed — Physician Decision | 2 | 1
Not completed — Move from study area | 3 | 2
Not completed — To militarycamp for conscript | 1 | 0
Not completed — To drug therapy course | 0 | 1
Not completed — Move to work oversea | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine | Total
Number analyzed (Participants) | 630 | 315 | 945
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.26 (9.40) | 29.32 (9.34) | 29.28 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 180 | 541
  Male | 269 | 135 | 404
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Thais | 630 | 315 | 945
Region of Enrollment [Count of Participants; unit: Participants] — Participants all Thais with age 18-49 years old on the day of screening and having Thai ID card or equivalent
  Participants
    Thailand | 630 | 315 | 945

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Seroconverted Participants at 21 Days Post-vaccination
Description: Seroconversion is defined as a serum HI antibody titer meeting the following four fold rising criteria.
  Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 21 of ≥1:40; or Pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination measured on Day 21.
  Measured against each of the 3 antigens
Time Frame: pre-vaccination (Day 0), 21 days post-vaccination
Population: Seroconversion against the hemagglutinin antigens contained in the vaccine were assessed in all studied participants. The analysis was performed as intention-to-treat (ITT).
Measure: Count of Participants; unit: Participants
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
Number analyzed (Participants) | 630 | 315
Participants
  Seroconversion Flu A H1 at Day 21 | 413 | 216
  Seroconversion Flu A H3 at Day 21 | 411 | 201
  Seroconversion Flu B at Day 21 | 425 | 199

2. Primary Outcome: Geometric Mean Titers (GMTs) of Participants at 21 Days Post-vaccination
Description: Geometric mean titers (GMTs) of serum HI antibodies pre- (Day 0) and post-vaccination (Day 21) for each of the three vaccine antigens.
  Note that titers below the lowest limit of quantitation (i.e., below the starting dilution of assay reported as "< 10") will be set to half that limit (i.e., 10/ 2 = 5). If a titer is reported as greater or equal to the upper limit of the assay, it will be set to that limit.
Time Frame: pre-vaccination (Day 0), 21 days post-vaccination
Population: Geometric mean titer against the hemagglutinin antigens contained in the vaccine were assessed in all studied participants. The analysis was performed as intention-to-treat (ITT).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
Number analyzed (Participants) | 630 | 315
titer
  GMT Flu A H1 at Day 0 | 40.67 [36.46 to 45.36] | 42.82 [36.78 to 49.86]
  GMT Flu A H1 at Day 21 | 326.09 [300.10 to 354.34] | 459.64 [405.05 to 521.59]
  GMT Flu A H3 at Day 0 | 45.55 [41.04 to 50.54] | 45.35 [39.09 to 52.60]
  GMT Flu A H3 at Day 21 | 349.30 [317.79 to 383.93] | 297.38 [261.48 to 338.21]
  GMT Flu B at Day 0 | 18.00 [16.27 to 19.90] | 19.27 [16.71 to 22.21]
  GMT Flu B at Day 21 | 165.96 [151.37 to 181.97] | 139.72 [123.23 to 158.42]

3. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events Post-vaccination.
Description: Solicited local and systemic adverse events within 30 minutes of vaccination and over the 3-day period post vaccination.
  Percentage of participants experiencing each reaction was calculated. Analysis based on Intention to Treat analysis
Time Frame: 30-minutes period,day 1,day 2 and day 3 post-vaccination period
Population: The analysis was conducted for participants who were randomized and received a study vaccination. Analysis based on Intention to Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
Number analyzed (Participants) | 630 | 315
Participants
  Pain, 30 min | 115 | 30
  Pain, Day 1 | 144 | 88
  Pain, Day 2 | 38 | 28
  Pain,Day 3 | 7 | 6
  Limitation of arm movement, 30 min | 52 | 14
  Limitation of arm movement, Day 1 | 64 | 25
  Limitation of arm movement, Day 2 | 11 | 10
  Limitation of arm movement, Day 3 | 2 | 2
  Headache, 30 min | 6 | 3
  Headache, Day 1 | 42 | 20
  Headache, Day 2 | 25 | 12
  Headache, Day 3 | 11 | 3
  Fatigue, 30 min | 8 | 4
  Fatigue, Day 1 | 60 | 36
  Fatigue, Day 2 | 26 | 15
  Fatigue, Day 3 | 16 | 6
  Malaise, 30 min | 4 | 3
  Malaise, Day 1 | 50 | 24
  Malaise, Day 2 | 20 | 7
  Malaise, Day 3 | 17 | 4
  Chills, 30 min | 4 | 3
  Chills, Day 1 | 12 | 4
  Chills, Day 2 | 7 | 1
  Chills, Day 3 | 4 | 1
  Myalgia, 30 min | 11 | 12
  Myalgia, Day 1 | 61 | 34
  Myalgia, Day 2 | 23 | 16
  Myalgia, Day 3 | 15 | 8
  Arthralgia, 30 min | 5 | 4
  Arthralgia, Day 1 | 18 | 10
  Arthralgia, Day 2 | 11 | 3
  Arthralgia, Day 3 | 5 | 0
  Nausea, 30 min | 1 | 2
  Nausea, Day 1 | 6 | 3
  Nausea, Day 2 | 4 | 2
  Nausea, Day 3 | 1 | 0
  Vomiting, 30 min | 0 | 0
  Vomiting, Day 1 | 0 | 1
  Vomiting, Day 2 | 1 | 1
  Vomiting, Day 3 | 1 | 0
  Rash, 30 min | 0 | 0
  Rash, Day 1 | 5 | 1
  Rash, Day 2 | 6 | 0
  Rash, Day 3 | 2 | 0

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events.
Description: Unsolicited adverse events (AEs) occurring within 90 days post-vaccination. Percentage of participants experiencing each reaction will be calculated.
Time Frame: within 90 days post-vaccination
Population: The analysis was conducted for participants who were randomized and received a study vaccination by Intention to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
Number analyzed (Participants) | 630 | 315
Participants
  Influenza like Illness (ILI) | 7 | 3
  Pyrexia | 24 | 12
  Influenza | 2 | 0
  Pharyngitis | 4 | 1
  Tonsillitis | 4 | 0
  Tonsillitis bacterial | 1 | 0
  Upper respiratory tract infection | 111 | 44
  Arthralgia | 1 | 0
  Myalgia | 5 | 3
  Dizziness | 4 | 0
  Headache | 40 | 16
  Cough | 12 | 4
  Productive cough | 2 | 0
  Rhinitis | 5 | 2
  Rhinorrhoea | 27 | 6
  Sneezing | 1 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | GPO Tri Fluvac Vaccine | Licensed Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/630 | 1/315
Serious Adverse Events (participants affected / at risk) | 1/630 | 1/315
Other Adverse Events (participants affected / at risk) | 273/630 | 114/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPO Tri Fluvac Vaccine (N=630) | Licensed Influenza Vaccine (N=315)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — FRACTURE LATERAL MAXILLARY SINUS AND LEFT ORBIT DUE TO MOTORCYCLE ACCIDENT
myocardial hypertrophy with infarction (Cardiac disorders) | 0 (0) | 1 (1) — myocardial hypertrophy with infarction
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPO Tri Fluvac Vaccine (N=630) | Licensed Influenza Vaccine (N=315)
Pyrexia (General disorders) | 24 (24) | 12 (13)
upper respiratory tract infection (Infections and infestations) | 111 (118) | 44 (47)
headache (Nervous system disorders) | 40 (44) | 16 (20)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 6 (6)
adominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 4 (4)
Toothache (Gastrointestinal disorders) | 5 (5) | 3 (3)
Influenza like illness (General disorders) | 7 (7) | 3 (3)
pharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
dysmenorrhoea (Reproductive system and breast disorders) | 6 (8) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 4 (4)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03390166/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03390166/SAP_001.pdf